CLINICAL TRIAL: NCT05865171
Title: A Phase 1, Open-label Study Evaluating the Pharmacokinetics and Safety of a Single Dose of Inaxaplin in Subjects With Severe Renal Impairment and Healthy Subjects With Normal Renal Function
Brief Title: A Study to Evaluate Pharmacokinetics (PK) and Safety of Inaxaplin in Participants With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: VX19-147-007
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Severe Renal Impairment (Experimental): Participants will receive a single dose of IXP on Day 1.
  Interventions: Drug: IXP
- Cohort 1: Healthy Participants (Experimental): Participants will receive a single dose of IXP on Day 1.
  Interventions: Drug: IXP

INTERVENTIONS:
Drug: IXP — Tablets for oral administration.
  Other Names: VX-147; Inaxaplin

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of a single dose of Inaxaplin (IXP) in participants with severe renal impairment and healthy participants with normal renal function.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.5 to 40.0 kilogram per meter square (kg/m^2)
* Stable renal function for at least 1 month prior to enrollment

Key Exclusion Criteria:

* Uncontrolled hypertension
* Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of IXP | Day 1 up to Day 7
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of IXP | Day 1 up to Day 7

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse events (AEs) and Serious Adverse Events (SAEs) | Day 1 through completion of study participation (up to a maximum of 17 days)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GCP Research, Ocala, Florida
  - Genesis Clinical Research, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing